CLINICAL TRIAL: NCT06634888
Title: Root Resorption and Alveolar Bone in the Maxillary Canine Retraction Using Injectable Platelet-rich Fibrin: A Split-Mouth Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PhamThiMinhChauCtump
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2022-07

CONDITIONS: Angle Class I
Keywords: injectable platelet-rich fibrin; canine retraction; root resorption
MeSH Terms: conditions — Malocclusion, Angle Class I; Root Resorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right sides were randomly allocated to treatments with i-PRF (Experimental): The amount of i-PRF was standardized as 2mL and was injected submucosal into the distobuccal and distopalatal side of the canine tooth (1mL for each side) under local anesthesia for pain control.
  Interventions: Diagnostic Test: Injectable platelet rich fbirin
- Left sides were randomly allocated to control sides. (Placebo Comparator): The placebo was standardized as 2mL and was injected submucosal into the distobuccal and distopalatal side of the canine tooth (1mL for each side) under local anesthesia for pain control.
  Interventions: Diagnostic Test: Injectable platelet rich fbirin

INTERVENTIONS:
Diagnostic Test: Injectable platelet rich fbirin — After the leveling and alignment phase, the canines were retracted with 150gm forces. The i-PRF was prepared from the blood of each patient then injected immediately before canine retraction on the buccal and palatal aspects of the extraction sites. All patients in this study were submitted for Cone beam computed tomography (CBCT) scanning before and after canine retraction. Cone beam computed tomography (CBCT) was used before and four months after retraction, with imaging conducted using the Orthophos SL 3D X-ray machine (Dentsply Sirona, Charlotte, CA, USA) while adhering to As Low As Reasonably Achievable (ALARA) guidelines to minimize radiation exposure
  Arms: Right sides were randomly allocated to treatments with i-PRF
Diagnostic Test: Injectable platelet rich fbirin — All patients in this study were submitted for Cone beam computed tomography (CBCT) scanning before and after canine retraction. Cone beam computed tomography (CBCT) was used before and four months after retraction, with imaging conducted using the Orthophos SL 3D X-ray machine (Dentsply Sirona, Charlotte, CA, USA) while adhering to As Low As Reasonably Achievable (ALARA) guidelines to minimize radiation exposure
  Arms: Left sides were randomly allocated to control sides.

SUMMARY:
Prolonged orthodontic treatment is a risk factor for root resorption, so accelerating the speed of tooth movement using different methods can limit tooth root resorption. There are multiple factors causing root resorption, such as orthodontic force level, treatment duration, and methods of quantification of root resorption. PRF, a completely autologous fibrin matrix, was developed as a second-generation platelet concentrate without adding anticoagulants and additives. The injectable platelet-rich fibrin is the liquid form of the substance obtained through low-speed centrifugation. It has many advantages over the conventional form, such as higher rates of regenerative cells and growth factors. In the present study, Cone Beam Computed Tomography (CBCT) was used as a measurement tool for root resorption. CBCT is a helpful tool for evaluating changes in the root length of teeth and surrounding bone tissue.

DETAILED DESCRIPTION:
Orthodontic treatment encompasses not only the correction of malocclusion and enhancement of dental arch aesthetics but also the preservation or restoration of optimal function and periodontal tissue health. Orthodontic tooth movement (OTM) is stimulated by remodeling the periodontal ligament (PDL) and alveolar bone. Bone remodeling is a process of both bone resorption on the pressure side and bone formation on the tension site.

Prolonged orthodontic treatment is a risk factor for root resorption, so accelerating the speed of tooth movement using different methods can limit tooth root resorption. Root resorption is an undesirable effect that occurs during orthodontic treatment. It is defined as a reduction of root length or cringe. Because root resorption is a multifactorial issue, it is essential to know and focus on the controlling factors that cause root resorption. Therefore, attempts to accelerate tooth movement and reduce treatment duration are significant to orthodontists and patients. Adequate alveolar bone volume and root length are prerequisite conditions for successful orthodontic tooth movement and post-treatment stability orthodontic tooth movement causes the inflammatory process in the periodontium to occur.

Platelet-based preparations from the patient's blood provide a safe alternative to commercially available bioactive materials. PRF, a completely autologous fibrin matrix, was developed as a second-generation platelet concentrate without adding anticoagulants and additives. The injectable platelet-rich fibrin (i-PRF) is the liquid form of the substance that is obtained through low-speed centrifugation (700rpm in 3 minutes) and has many advantages over the conventional form, such as higher rates of regenerative cells and growth factors such as prostaglandins, interleukins, the tumor necrosis factor-a superfamily, and receptor activator of nuclear factor (RANK)/RANK ligand (RANKL)/osteoprotegerin (OPG) are increased in the PDL during orthodontic tooth movement . The presence of these inflammatory mediators in the PDL during orthodontic tooth movement indicates their role in the occurrence of orthodontically induced tooth root resorption.

Cone beam computed tomography (CBCT) imaging allows for a three-dimensional evaluation of teeth and their adjacent anatomical structures, resulting in a detailed visualization of the tooth and its neighboring structures. Subsequently, the area of the tooth resorption can be detected easily. CBCT imaging allows radiation to be focused on the area of anatomical interest while encompassing all hard and soft tissues in three dimensions, providing more significant information with a potential decrease in cumulative radiation exposure for patients.

Little is known about the effects of the placement of these biomaterials on the root length of the moved tooth and on the surrounding supporting bone tissue during orthodontic movement. This study aimed to evaluate and compare these effects after distalization of maxillary canines in alveolar preserved with i-PRF and control alveolar in adult patients using Cone beam computed tomography (CBCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed long-term tooth replacement have cervical vertebral maturity at stages CS5, CS6 according to the classification of Baccetti et al.
* Patients with type I Angle malformation have bilateral maxillary first small canines
* No missing teeth except third molars
* No previous orthodontic treatment
* Absence of systemic diseases and dentofacial anomalies, had good periodontal health, had typical values of blood tests, e.g., bleeding time 1 - 4 minutes, coagulation time 5 - 10 minutes
* Patients agreed to participate in the study.

Exclusion Criteria:

* Patients suffering from bleeding disorders, diabetes, bone diseases, periodontal disease, and cancer are using drugs such as aspirin, heparin, warfarin, non-steroidal anti-inflammatory drugs, and glucocorticoids... affects the speed of tooth movement and the ability to clot and stop bleeding.
* The patient has trauma and facial deformities
* The patient smokes and is pregnant. The patient had other teeth extracted except the first premolar

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-27 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Our study aims to investigate the effectiveness of i-PRF in root resorption | Our study aims to investigate the effectiveness of i-PRF in root resorption using On Demand 3D software at the time before and 4 months after canine distalization (T0) & (T4)
  CBCT was used before (T0) and four months (T4) after retraction, with imaging conducted using On Demand 3D software according to the As Low As Reasonably Achievable guidelines.

SECONDARY OUTCOMES:
Our study aims to investigate the effectiveness of i-PRF in alveolar bone density. | Our study aims to investigate the effectiveness of i-PRF in alveolar bone density using On Demand 3D software at the time before and 4 months after canine distalization (T0) & (T4)
  CBCT was used before (T0) and four months (T4) after retraction, with imaging conducted using On Demand 3D software according to the As Low As Reasonably Achievable guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Can Tho University of Medicine and Pharmacy, Can Tho, Vietnam

REFERENCES:
- [Result] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Three-dimensional evaluation of the effects of injectable platelet rich fibrin (i-PRF) on alveolar bone and root length during orthodontic treatment: a randomized split mouth trial. BMC Oral Health. 2021 Mar 2;21(1):92. doi: 10.1186/s12903-021-01456-9. PMID 33653326